CLINICAL TRIAL: NCT02960022
Title: A Phase 2 Open-label Extension Study for Subjects With Prostate Cancer Who Previously Participated in an Enzalutamide Clinical Study
Brief Title: A Study for Subjects With Prostate Cancer Who Previously Participated in an Enzalutamide Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0123; 2016-001694-32 (EudraCT Number); 2023-510298-33-00 (Registry Identifier: EU CTIS); jRCT2031220674 (Registry Identifier: jRCT)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prednisone; MDV3100; enzalutamide; Xtandi; abiraterone acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Abiraterone Acetate; Prednisone; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- enzalutamide (Experimental): Subjects will receive enzalutamide orally once daily at the same time each day
  Interventions: Drug: enzalutamide
- enzalutamide plus abiraterone acetate and prednisone (Experimental): Subjects enrolling from study 9785-CL-0011 or MDV3100-10 (PLATO) study may receive abiraterone acetate once daily and prednisone twice daily, in addition to enzalutamide once daily
  Interventions: Drug: enzalutamide; Drug: abiraterone acetate; Drug: prednisone
- Enzalutamide plus leuprolide acetate (Experimental): Subjects enrolling from study MDV3100-13 (EMBARK) study may receive leuprolide acetate once every 12 weeks in addition to enzalutamide once daily
  Interventions: Drug: enzalutamide; Drug: Leuprolide acetate

INTERVENTIONS:
Drug: enzalutamide — Subjects will receive enzalutamide orally once daily at the same time each day.
  Other Names: MDV3100; Xtandi
Drug: abiraterone acetate — Subjects enrolling from study 9785-CL-0011 or MDV3100-10 (PLATO) study may receive abiraterone acetate once daily and prednisone twice daily, in addition to enzalutamide
  Arms: enzalutamide plus abiraterone acetate and prednisone
Drug: prednisone — Subjects enrolling from study 9785-CL-0011 or MDV3100-10 (PLATO) study may receive abiraterone acetate once daily and prednisone twice daily, in addition to enzalutamide
  Arms: enzalutamide plus abiraterone acetate and prednisone
Drug: Leuprolide acetate — Subjects enrolling from study MDV3100-13 (EMBARK) study may receive leuprolide acetate once every 12 weeks in addition to enzalutamide once daily
  Arms: Enzalutamide plus leuprolide acetate

SUMMARY:
The purpose of this study is to collect long term safety data in subjects who are continuing to derive clinical benefit from treatment with Enzalutamide from the subjects participation in an enzalutamide clinical study sponsored by Astellas or Medivation (i.e., parent study) which has completed, at a minimum, the primary analysis or the study specified evaluation period.

DETAILED DESCRIPTION:
Subjects must continue on the treatment regimen that the subject was receiving in the prior study. Dose changes of any of the prior therapies subjects were receiving on the previous protocol are allowed after medical monitor approval. The day 1 visit for this study should coincide with the last treatment visit for the study the subject will be enrolling from (≤ 7 days post last visit of parent study). The subjects will be followed according to the local institution's standard of care and will be required to return to the institution every 24 weeks (± 7 days) to review adverse events (AEs), collect concomitant medications and confirm that no discontinuation criteria are met. At each visit and at every 12 weeks (IP only visit) subjects are to return all dispensed study drug and to receive more study drug if applicable. All AEs (new and ongoing from the study the subject is enrolling from) and Serious Adverse Events (SAEs) (including death), will be collected from the time the subject signs the consent form until the end of study visit.

After the marketing approval in South Korea, this study continued as "post marketing clinical study" in South Korea. In the rest of the countries which participated in this study, this study continued as clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must currently be receiving enzalutamide for prostate cancer in a study sponsored by Astellas or Medivation and, based on the investigator's assessment, benefit from continued treatment. Subjects participating in investigator-initiated trials are not eligible.
* Subject is able to continue on the treatment regimen that the subject was receiving in the prior study. If in the investigator's assessment, a change is needed to the subject's regimen (e.g., dose change in Androgen deprivation therapy (ADT) or dropping of a combination therapy) approval from a medical monitor is required prior to enrollment.
* Subject is able to swallow enzalutamide capsules and comply with study requirements.
* Subject and female partner who is of childbearing potential must continue to use 2 forms of birth control, of which 1 must be highly effective and 1 must be a barrier method throughout the study and for 3 months after final enzalutamide administration.
* Subject agrees to avoid sperm donation during the study and for at least 3 months after final enzalutamide administration.
* Subject agrees not to participate in another interventional study while on treatment.

Canada Specific:

* Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization for the United States sites) must be obtained from the subject prior to any study-related procedures.
* Subject must currently be receiving enzalutamide for breast cancer in a study sponsored by Astellas or Medivation/Pfizer and based on the investigator's assessment, benefit from continued treatment. Subjects participating in investigator-initiated trials are not eligible.
* Subject is able to continue on the treatment regimen that they were receiving in the prior study. If in the investigator's assessment, a change is needed to the subject's regimen (e.g., dropping of a combination therapy) approval from a medical monitor is required prior to enrollment.
* Subject is able to swallow enzalutamide capsules and comply with study requirements.
* Subject is either:
* Of nonchildbearing potential:
* postmenopausal (defined as no spontaneous menses for at least 12 months prior to Day 1 with follicle stimulating hormone (FSH) > 40 IU/L at Day 1 for women < 55 years of age),
* documented surgically sterile or status post hysterectomy (at least 1 month prior to Day 1),
* Or, if of childbearing potential,
* must have a negative urine pregnancy test at Day 1 before the first dose of study drug is administered,
* must use 2 acceptable methods of birth control starting at Day 1 and through 6 months after the final study drug administration,
* must not donate ova starting at first administration of study intervention and throughout 6 months after final study intervention administration.

The 2 acceptable methods of birth control are as follows or per local guidelines where these require additional description of contraceptive methods:

* A barrier method (e.g., condom by a male partner) is required; AND
* One of the following is required:
* Placement of an intrauterine device (IUD) or intrauterine system (IUS);
* Additional barrier method including occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository;
* Vasectomy or other surgical castration at least 6 months before Day 1.
* The subject must not be breastfeeding at Day 1 or during the study period, and for 6 months after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject met any of the discontinuation criteria or whose cancer progressed on the current enzalutamide clinical study in which subject is enrolling from.
* Subject requires treatment with or plans to use either of the following:

  * New systemic therapy for subjects cancer (palliative radiation therapy is allowed). The treatment with agents administered during previous studies which was stopped and then restarted during this study does not represent new treatment.
  * Investigational therapy other than enzalutamide.
* Subject is currently participating in an investigator-initiated interventional trial and receiving enzalutamide.
* Subject has any concurrent disease, infection, or comorbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data.

Canada Specific:

Subject will be excluded from participation if any of the following apply:

* Subject met any of the discontinuation criteria or whose cancer progressed on the current enzalutamide clinical study in which they are enrolling from.
* Subject requires treatment with or plans to use any of the following:
* New systemic therapy for their cancer (palliative radiation therapy is allowed). The treatment with agents administered during previous studies which was stopped and then restarted during this study does not represent new treatment.
* Investigational therapy other than enzalutamide.
* Subject is currently participating in an investigator-initiated interventional trial and receiving enzalutamide.
* Subject has any concurrent disease, infection, or comorbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2016-12-22 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Until End of Study (Up to 96 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (241):
- United States (50):
  - Site US10052, Anchorage, Alaska
  - Site US10011, Tucson, Arizona
  - Site US10040, Los Angeles, California
  - Site US10009, Los Angeles, California
  - Site US10067, Orange, California
  - Site US10008, San Bernardino, California
  - Site US10042, San Diego, California
  - Site US10028, Stanford, California
  - Site US10001, Aurora, Colorado
  - Site US10017, Denver, Colorado
  - Site US10050, Washington D.C., District of Columbia
  - Site US10049, Daytona Beach, Florida
  - Site US10048, Jacksonville, Florida
  - Site US10002, Chicago, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Site US10007, Jeffersonville, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Site US10066, Lenexa, Kansas
  - Site US10029, Towson, Maryland
  - Site US10032, St Louis, Missouri
  - Nebraska Medical Hospital, Omaha, Nebraska
  - Site US10023, Omaha, Nebraska
  - Site US10004, Hackensack, New Jersey
  - Site US10024, Garden City, New York
  - Site US10055, New York, New York
  - Site US10059, New York, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - Site US10053, Syracuse, New York
  - Site US10030, Chapel Hill, North Carolina
  - Site US10062, Charlotte, North Carolina
  - Site US10020, Concord, North Carolina
  - Site US10031, Greensboro, North Carolina
  - Eastern Urological Associates, Greenville, North Carolina
  - Site US10046, Winston-Salem, North Carolina
  - Site US10035, Cincinnati, Ohio
  - Site US10022, Springfield, Oregon
  - Site US10027, Lancaster, Pennsylvania
  - Site US10005, Pittsburgh, Pennsylvania
  - Site US10018, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Site US10003, Myrtle Beach, South Carolina
  - Site US10041, Nashville, Tennessee
  - Site US10010, Dallas, Texas
  - Site US10034, Houston, Texas
  - Site US10043, Houston, Texas
  - Site US10014, Norfolk, Virginia
  - Site US10015, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Site US10038, Seattle, Washington
  - Site US10021, Madison, Wisconsin
- Argentina (6):
  - Site AR54005, Buenos Aires, Buenos Aires F.D.
  - Site AR54007, Rosario, Santa Fe Province
  - Site AR54008, Buenos Aires
  - Site AR54003, Cordorba
  - Site AR54006, San Miguel de Tucumán
  - Site AR54002, San Miguel de Tucumán
- Australia (12):
  - Site AU61014, Albury, New South Wales
  - Site AU61001, Tweed Heads, New South Wales
  - Site AU61012, Wahroonga, New South Wales
  - Site AU61017, Wahroonga, New South Wales
  - Site AU61006, Ashford
  - Site AU61019, Ballarat
  - Site AU61007, East Bentleigh
  - Site AU61009, Malvern
  - Site AU61021, Parkville
  - Site AU61008, South Brisbane
  - Site AU61016, St Albans
  - Site AU61004, Westmead
- Site AT43001, Vienna, Austria
- Belgium (9):
  - Site BE32002, Kortrijk, West-Vlaanderen
  - Site BE32009, Anderlecht
  - Site BE32004, Brussels
  - Site BE32005, Ghent
  - Site BE32011, Ghent
  - Site BE32007, Hasselt
  - Site BE32008, Leuven
  - Site BE32001, Liège
  - Site BE32003, Turnhout
- Brazil (7):
  - Site BR55007, Porto Alegre, Rio Grande do Sul
  - Site BR55009, Bahia
  - Site BR55008, Campinas
  - Site BR55004, Ijuí
  - Site BR55011, Jaú
  - Site BR55002, Rio Grande
  - Site BR55010, Santo André
- Canada (8):
  - Site CA15003, Kingston, Ontario
  - Site CA15021, Toronto, Ontario
  - Site CA15001, Granby, Quebec
  - Site CA15019, Abbotsford
  - Site CA15020, Greenville
  - Site CA15011, Montreal
  - Site CA15017, Oakville
  - Site CA15022, Québec
- Chile (6):
  - Site CL56006, Viña del Mar, Región de Valparaíso
  - Site CL56007, Santiago, RM
  - Site CL56005, Santiago, RM
  - Site CL56004, IX Region
  - Site CL56002, Santiago
  - Site CL56001, Viña del Mar
- China (3):
  - Site CN86003, Hubei
  - Site CN86010, Hunan
  - Site CN86005, Nanjing
- Czechia (4):
  - Site CZ42004, Olomouc
  - Site CZ42002, Olomouc
  - Site CZ42001, Prague
  - Site CZ42003, Prague
- Denmark (5):
  - Site DK45002, Aalborg, North Denmark
  - Site DK45003, Aarhus
  - Site DK45001, Copenhagen
  - Site DK45004, Herlev
  - Site DK45006, Vejle
- Finland (2):
  - Site FL35802, Tampere
  - Site FL35805, Turku
- France (12):
  - Site FR33021, Bordeaux
  - Site FR33008, La Roche-sur-Yon
  - Site FR33010, Lille
  - Site FR33002, Lyon
  - Site FR33020, Montpellier
  - Site FR33006, Nîmes
  - Site FR33003, Paris
  - Site FR33017, Paris
  - Site FR33001, Saint-Herblain
  - Site FR33019, Strasbourg
  - Site FR33022, Strasbourg
  - Site FR33004, Villejuif
- Site GE99501, Tbilisi, Georgia
- Germany (7):
  - Site DE49004, Nürtingen, Baden-Wurttemberg
  - Site DE49007, Waldshut-Tiengen, Baden-Wurttemberg
  - Site DE49006, Mannheim, DE
  - Site DE49001, Duisburg, North Rhine-Westphalia
  - Site DE49010, Bonn
  - Site DE49003, Hamburg
  - Site DE49013, Hamburg
- Site HK85202, Hong Kong, Hong Kong
- Israel (5):
  - Site IL97206, Haifa
  - Site IL97205, Jerusalem
  - Site IL97202, Peth Tikva
  - Site IL97204, Ramat Gan
  - Site IL97203, Tzrifin Beer Yakov
- Italy (8):
  - Site IT39008, Faenza (RA), Emilia-Romagna
  - Site IT39001, Arezzo
  - Site IT39011, Candiolo
  - Site IT39004, Cremona
  - Site IT39002, Forlì
  - Site IT39005, Roma
  - Site IT39009, Toscana
  - Site IT39006, Trento
- Japan (14):
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Kyushu University Hospital, Higashiku, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Kagawa University Hospital, Kida-gun, Kagawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koutou-ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba cancer center, Chiba
  - Harasanshin hospital, Fukuoka
  - Kyoto University hospital, Kyoto
  - Niigata University Medical and Dental Hospital, Niigata
  - Osaka Metropolitan University Hospital, Osaka
- Site MY60001, Kuching, Malaysia
- Site MD37301, Chisinau, Moldova
- Netherlands (4):
  - Site NL31010, Amsterdam
  - Site NL31009, Den Helder
  - Site NL31004, Maastricht
  - Site NL31011, Rotterdam
- New Zealand (3):
  - Site NZ64002, Auckland
  - Site NZ64005, Dunedin
  - Site NZ64001, Hamilton
- Site NO47001, Stavanger, Norway
- Poland (6):
  - Site PL48002, Gdansk
  - Site PL48001, Mysłowice
  - Site PL48004, Pozman
  - Site PL48005, Słupsk
  - Site PL48011, Warsaw
  - Site PL48003, Wroclaw
- Romania (3):
  - Site RO40003, Bucharest
  - Site RO40001, Cluj-Napoca
  - Site RO40004, Cluj-Napoca
- Russia (6):
  - Site RU70008, Ivanovo
  - Site RU70001, Moscow
  - Site RU70005, Omsk
  - Site RU70009, Saint Petersburg
  - Site RU70003, Saint Petersburg
  - Site RU70006, Saint Petersburg
- Serbia (2):
  - Site RS38102, Belgrade
  - Site RS38101, Belgrade
- Slovakia (7):
  - Site SK10223, Bratislava
  - Site SK42109, Košice
  - Site SK42106, Košice
  - Site SK42105, Nitra
  - Site SK42103, Prešov
  - Site SK42108, Trenčín
  - Site SK42107, Žilina
- Site ZA27001, George, South Africa
- South Korea (10):
  - Site KR82008, Busan
  - Site KR82012, Seongnam-si
  - Site KR82005, Seongnam-si
  - Site KR82009, Seoul
  - Site KR82007, Seoul
  - Site KR82011, Seoul
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82003, Seoul
  - Site KR82004, Seoul
- Spain (10):
  - Site ES34007, Barcelona
  - Site ES34003, Barcelona
  - Site ES34004, Barcelona
  - Site ES34011, Girona
  - Site ES34012, Madrid
  - Site ES34001, Madrid
  - Site ES34008, Madrid
  - Site ES34005, Pamplona
  - Site ES34014, Salamanca
  - Site ES34010, Santiago de Compostela
- Sweden (2):
  - Site SE46001, Gothenburg
  - Site SE46003, Umeå
- Taiwan (5):
  - Site TW88607, Guishan
  - Site TW88603, Kaohsiung City
  - Site TW88601, Kaohsiung City
  - Site TW88602, Taichung
  - Site TW88606, Taipei
- Thailand (2):
  - Site TH66001, Hat Yai, Changwat Songkhla
  - Site TH66002, Bangkok
- Site TR90002, Beşevler, Ankara, Turkey (Türkiye)
- Ukraine (4):
  - Site UA38004, Dnipro
  - Site UA38005, Kharkiv
  - Site UA38001, Kyiv
  - Site UA38003, Uzhhorod
- United Kingdom (11):
  - Site GB44009, Bebington
  - Site GB44003, Belfast
  - Site GB44004, Bristol
  - Site GB44014, Cambridge
  - Site GB44005, Cardiff
  - Site GB44002, Glasgow
  - Site GB44006, London
  - Site GB44007, Manchester
  - Site GB44008, Northwood
  - Site GB44016, Nottingham
  - Site GB44001, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/